CLINICAL TRIAL: NCT03699319
Title: A Phase II/I Open-Label Clinical Trial of CPI-613 in Combination With Modified FOLFIRINOX in Patients With Locally Advanced Pancreatic Cancer and Good Performance Status
Brief Title: CPI-613 in Combination With Modified FOLFIRINOX in Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Bajor, MD (Other)
Responsible Party: Sponsor-Investigator, David Bajor, MD, MD, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2218
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Cancer
Keywords: FOLFIRINOX; CPI-613
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — devimistat; Oxaliplatin; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Intervention Model Description: Single-armed study of patients with locally advanced pancreatic cancer, evaluating combination CPI-613 with modified FOLFIRINOX
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Standard Dose Cohort: CPI-613 + mFOLFIRINOX (Experimental): Novel drug and mitochondrial inhibitor, CPI-613 in conjunction with standard-of-care FOLFRINOX.
  Consists of a Standard Dose Cohort and Dose escalation cohort using a standard 3 + 3 design starting at 750 mg/m^2 given at a rate of 4 ml/min ("dose level (DL) 2"). Participants receiving a dose of 1000mg/m^2 will be treated over 2 hours. In the absence of any DLT, the next DL will begin enrollment. If 1 DLT occurs, the DL will be expanded by 3 participants. If <33% of participants experience a DLT, the next DL will be opened and will proceed in similarly. Only 2 DLs are expected to be studied: 750 mg/m^2 and 1000 mg/m^2.
  Participants may be enrolled in this cohort after the accrual goal of the standard cohort is met but prior to the completion of treatment of all patients in the standard dose cohort
  Participants experiencing a DLT will be allowed to continue on the study at the standard DL of 500 mg or lower.
  Interventions: Drug: CPI 613; Drug: Oxaliplatin; Drug: Irinotecan; Drug: 5-flurouracil; Drug: Folinic acid

INTERVENTIONS:
Drug: CPI 613 — Standard Dose Cohort: CPI-613, 500 mg/m2, IV infusion at a rate of 4 mL/min via a central venous port on days 1 and 3 of each cycle, every 2 weeks.
  Dose Escalation Cohort: CPI-613, 750-1000 mg/m2 IV infusion at a rate of 3 mL/min via a central venous port on days 1 and 3 of each cycle, every 2 weeks.
  Intended treatment protocol is 12 cycles (2 weeks each) or 6 months
  Other Names: 6, 8-bis-benzylsulfanyloctanoic acid
Drug: Oxaliplatin — Administered at 65 mg/m2 given as a 2-hr IV
  Part of SOC mFOLFRINOX treatment combination of Oxaliplatin, Irniotecan, 5-flurouracil, and vitamin derivative (Folinic acid)
  Other Names: Eloxatin
Drug: Irinotecan — Administered at 140 mg/m2 given as a 90-min IV infusion) via a Y-connector
  Part of SOC mFOLFRINOX treatment combination of Oxaliplatin, Irniotecan, 5-flurouracil, and vitamin derivative (Folinic acid)
  Other Names: Camptosar
Drug: 5-flurouracil — Administered at 400 mg/m2 as bolus followed by a 46-hr infusion at 2400 mg/m2, starting immediately after completion of folinic acid and irinotecan
  Part of SOC mFOLFRINOX treatment combination of Oxaliplatin, Irniotecan, 5-flurouracil, and vitamin derivative (Folinic acid)
  Other Names: 5FU
Drug: Folinic acid — Administered at 400 mg/m2 given as a 90-min infusion immediately after oxaliplatin
  Part of SOC mFOLFRINOX treatment combination of Oxaliplatin, Irniotecan, 5-flurouracil, and vitamin derivative (Folinic acid)
  Other Names: Leucovorin; Calcium folinate; FA

SUMMARY:
The purpose of this study is to treat participants with the combination of CPI-613 (the study drug) with FOLFIRINOX (the standard combination of drugs) to determine if it is safe and effective for participants with localized and unresectable pancreatic cancer. This study is specifically for participants who have a pancreatic cancer that is localized and not considered resectable or removable by a surgeon, without additional treatment.

DETAILED DESCRIPTION:
This is a single-arm study of participants with locally advanced pancreatic ductal adenocarcinoma evaluating combination CPI-613 with modified FOLFIRINOX, with the addition of a dose escalation cohort to assess safety. All study participants will get the same study intervention, which includes the best available treatment for locally advanced pancreatic cancer, plus an experimental therapy. The standard therapy is called mFOLFIRINOX, which is a combination of three chemotherapy drugs (Oxaliplatin, Irniotecan and 5-flurouracil) and one additional vitamin derivative (Folinic acid). The experimental drug is CPI-613, which inhibits energy production in cells, and early studies suggest that pancreatic cancer cells may be especially sensitive. Pre-treatment, diagnostic biopsy tissue will be collected when available, and clinical data will be evaluated to determine if the combination results in improved overall survival compared to historical experience. Based on new data, the study team will also attempt to identify a new maximum tolerated dose (MTD) of CPI-613 in a phase 1 open-label dose-regimen finding study.

The objectives of the Standard Dose Cohort are to determine the safety and efficacy of CPI-613, in combination with mFOLFIRINOX for locally advanced pancreatic cancer.

The objectives of the Dose Escalation Cohort is to determine a new maximum-tolerated dose (MTD) of CPI-613 when given in combination with mFOLFIRINOX.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed pancreatic adenocarcinoma.
* Participants must have locally advanced (including unresectable or borderline resectable) pancreatic cancer based on CT or MRI imaging (pancreas protocol CT of the abdomen and pelvis if possible, MRI with contrast or CT with oral and IV contrast in the absence of a pancreas protocol CT scan, CT of the chest with or without contrast) as determined by the PI or Co-investigators. Participants with contrast allergies may be permitted without contrast scans if approved by the PI or Co-Investigators for safety reasons.
* Eastern Cooperative Oncology Group (ECOG) Performance status being 01 within 1 week of planned start of therapy.
* Participants must have normal organ and marrow function as defined below < 2 weeks must be:

  * Adequate hematologic (white blood cell [WBC] >= 3500 cells/mm3; platelet count >= 100,000 cells/mm3; absolute neutrophil count [ANC] >=1500 cells/mm3; and hemoglobin >=8 g/dL).
  * Adequate hepatic function (aspartate aminotransferase [AST/SGOT] 3x upper normal limit [UNL], alanine aminotransferase [ALT/SGPT] <=3x UNL, bilirubin <=1.5x UNL).
  * Adequate renal function (serum creatinine <=2.0 mg/dL or 177 µmol/L).
  * Adequate coagulation ("International Normalized Ratio" or INR must be <1.5) unless on therapeutic blood thinners.
* Expected survival >=3 months in the view of the PI or investigators.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation.
* Fertile men must practice effective contraceptive methods (i.e. surgical sterilization, or a condom used with a spermicide) during the study, unless documentation of infertility exists.
* No evidence of clinically significant active infection and no serious infection within the past month requiring hospitalization.
* Participants must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants with endocrine or acinar pancreatic carcinoma.
* Participants with resectable pancreatic cancer.
* Participants with metastatic pancreatic cancer based on imaging.
* Participants who have received prior surgical or medical treatment for pancreatic cancer.
* Participants receiving any other standard or investigational treatment for their cancer with a primary goal of improving survival within the past 2 weeks prior to initiation of CPI-613 treatment.
* Pregnant women or breast feeding women, or women of child-bearing potential not using reliable means of contraception are excluded from this study because the teratogenic or abortifacient effects of CPI-613 is unknown. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CPI-613, breastfeeding should be discontinued if the mother is treated with CPI-613. These potential risks may also apply to other agents used in this study.
* Fertile men unwilling to practice contraceptive methods during the study period.
* Participants with a life expectancy less than 3 months.
* Participants with a serious medical illness that would potentially increase participants' risk for toxicity
* Participants with any active uncontrolled bleeding, and any participnats with a bleeding diathesis (e.g., active peptic ulcer disease).
* Participants with a history of myocardial infarction that is <3 months prior to registration.
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure or coronary artery disease, unstable angina pectoris, cardiac arrhythmia, symptomatic myocardial infarction or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants who are known to be HIV-positive and on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with CPI-613.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Two years after completion of treatment
  Interval between enrollment and death for participants for all participants.
  Median OS will be estimated using the Kaplan-Meier method along with a two-sided 80% confidence interval (CI). OS will be documented and reported separately per cohort
MTD of CPI-613 when given in combination with mFOLFIRINOX | Up to 4 weeks from start of treatment
  MTD of CPI-613 when given in combination with mFOLFIRINOX in the added small cohort of participants with higher doses of CPI-613 developed to redefine MTD

SECONDARY OUTCOMES:
Median Progression free survival (PFS) | Two years after completion of treatment
  Median (and 95% CI) time from study enrollment to progression or death from any cause for all participants.
  Distribution of PFS will be estimated using the Kaplan-Meier method. Participants alive at the end of follow-up are censored. PFS will be documented and reported separately per cohort
Median Time to progression (TTP) | Two years after completion of treatment
  Median (and 95% CI) time from enrollment to progression
  Distribution of TTP will be estimated using the Kaplan-Meier method. Participants who die but have not progressed are censored.
Response rates per RECIST version 1.1 | Two years after completion of treatment
  RECIST version 1.1 response rates including complete response, partial response and stable disease (CR+PR+SD).
Complete pathologic response rates (CRp) | Two years after completion of treatment
  CRp defined as the proportion of participants that are designated having a complete response after treatment on protocol, evidenced by tissue samples taken during the subsequent resection
  CRp is defined by the NCI as "the lack of all signs of cancer in tissue samples removed during surgery or biopsy after treatment with radiation or chemotherapy".
Resection margins | Two years after completion of treatment
  Resection margins are defined by the NCI as "The edge or border of the tissue removed in cancer surgery. The margin is described as negative or clean when the pathologist finds no cancer cells at the edge of the tissue, suggesting that all of the cancer has been removed. The margin is described as positive or involved when the pathologist finds cancer cells at the edge of the tissue, suggesting that all of the cancer has not been removed."
  The rate of negative resection margins will be estimates with 95 % confidence intervals
Surgical resection rates | Up to 4 weeks from end of treatment
  Percent of participants previously determined to be borderline- or non-resectable that undergo complete surgical resection after treatment on protocol.

CONTACTS AND LOCATIONS:
Overall Officials: David Bajor, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States